CLINICAL TRIAL: NCT07106138
Title: Comparing the Effectiveness of Several Local Anaesthesic Systems and Thier Effect on Pain Anxiety Behaviour and Vital Signs in Children
Brief Title: Impact of Local Anesthesia Techniques on Children's Dental Treatment Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Tishreen U_pedodontic
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Dental Anxiety; Pain Management; Pediatric Dentistry
Keywords: Local anesthetic delivery systems; Computer-controlled anesthesia; Needle-free injection; Vibrotactile Devices; Dental anxiety; Pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional Syringe Group (Active Comparator): 28 Child received local anesthesia using a traditional dental syringe with standard technique.
  Interventions: Device: Conventional syringe injection
- CCLAD - Star Pen Group (Experimental): 28 Child received Local anesthesia using the Star Pen computer-controlled delivery system
  Interventions: Device: Star Pen
- Comfort-In - Needle-Free Group (Experimental): 28 Child received local anesthesia using the Comfort-In needle-free jet injector system.
  Interventions: Device: Comfort-In
- Vibraject - Vibrotactile Device Group (Experimental): 28 Child received Local anesthesia using a conventional syringe while applying the Vibraject vibrotactile stimulation device.
  Interventions: Device: Vibraject

INTERVENTIONS:
Device: Conventional syringe injection — Manual injection using a conventional dental syringe and needle to deliver local anesthetic.
  Arms: Conventional Syringe Group
Device: Star Pen — A computer-controlled local anesthetic delivery system designed to provide slow, controlled injection with improved comfort.
  Arms: CCLAD - Star Pen Group
Device: Comfort-In — A needle-free injection system that delivers anesthetic through high-pressure jet injection, reducing injection-related discomfort.
  Arms: Comfort-In - Needle-Free Group
Device: Vibraject — A vibrating attachment for dental syringes that provides vibrotactile stimulation during injection to distract from pain perception
  Arms: Vibraject - Vibrotactile Device Group

SUMMARY:
compare the effectiveness of several local anesthetic delivery systems in managing pain, anxiety, behavior, and vital signs among pediatric dental patients. A total of 112 children aged 6 to 10 years were included and randomly assigned to receive local anesthesia via one of the following methods: conventional syringe, computer-controlled local anesthetic delivery system (Star Pen), needle-free injector (Comfort-In), or a vibrotactile device (Vibraject). Pain was assessed using the FLACC and Wong-Baker FACES scales, anxiety with the Venham Picture Test, and behavior with the Houpt scale. Vital signs including pulse and oxygen saturation were recorded during treatment. Additionally, satisfaction levels of both the patients and their parents were evaluated using structured questionnaires and Likert scales. The study seeks to determine which technique provides the most comfortable and effective experience for children undergoing dental procedures.

DETAILED DESCRIPTION:
Local anesthesia is essential for pain control during pediatric dental procedures, yet its administration can cause significant anxiety and distress in children. Recent innovations aim to improve the delivery of anesthesia to make it less painful and more acceptable. This randomized clinical trial investigated and compared four local anesthetic systems: traditional syringe, computer-controlled local anesthetic delivery (CCLAD) using the Star Pen, needle-free injection using Comfort-In, and vibrotactile stimulation with Vibraject.

A total of 112 healthy children aged 6 to 10 years participated in the study. The children were randomly assigned to one of the four anesthesia groups. Pain perception was measured using both the FLACC scale and the Wong-Baker FACES Pain Rating Scale. Anxiety was evaluated using the Venham Picture Test before and during the procedure. Child behavior was rated using the Houpt Behavioral Scale. Vital signs including pulse rate and oxygen saturation were monitored at baseline and during treatment. In addition, satisfaction levels were assessed for both the pediatric patients and their accompanying parents, using child-friendly satisfaction questionnaires and parent-rated Likert scales.

This study aims to identify the anesthesia delivery method that best minimizes pain and anxiety, optimizes behavior, maintains physiological stability, and maximizes satisfaction, thereby enhancing the quality of care in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-10 years.
2. Physically healthy with no neurological disorders or systemic diseases.
3. Children classified as positive" or "negative-positive" according to the modified Frankl Behavioral Rating Scale.
4. Not taking any sedatives or analgesics drugs

Exclusion Criteria:

1. Uncooperative children who exhibit clear behavioral problems.
2. Children with systemic diseases or disorders that may interfere with local anesthesia.
3. Use of any medications that may affect vital signs or pain response.
4. Presence of infection at the injection site.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Pain level during dental anesthesia and treatment (behavioral assessment) | From the start of local anesthetic injection until completion of pulpotomy, assessed up to 30 minutes.
  Procedural pain was assessed using the FLACC scale, which evaluates five behavioral categories (Face, Legs, Activity, Cry, Consolability), each scored from 0 to 2, for a total score range of 0-10. Higher scores indicate greater pain.Scores were assigned by trained observers during the procedure.
Pain level during dental anesthesia and treatment (self-reported) | From the start of local anesthetic injection until completion of pulpotomy, assessed up to 30 minutes.
  Procedural pain was assessed using the Wong-Baker FACES Pain Rating Scale to measure children's self-reported pain, It's a self-reported scale with six cartoon faces representing increasing levels of pain, scored from 0 (no pain) to 10 (worst pain). Children were asked to point to the face that best described their pain.
  Higher scores on either scale indicated greater pain intensity.
Anxiety level during dental anesthesia and treatment | From the start of local anesthetic injection until completion of pulpotomy, assessed up to 30 minutes.
  Anxiety was measured using the Venham Picture Test (VPT),The test consists of eight pairs of cartoon images, each pair containing one figure showing a relaxed expression and one showing an anxious expression. Children were asked to choose the picture that best reflected how they felt. Scores ranged from 0 to 8, with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Child behavior during dental procedures | From the start of local anesthetic injection until completion of pulpotomy, assessed up to 30 minutes.
  Behavior was assessed using the Houpt Behavior Rating Scale, which evaluates cooperation during dental procedures.The scale is ranging from 1 (poor) to 6 (excellent). Higher scores indicated better cooperation and comfort during treatment.
Heart rate | From baseline measurement taken 5 minutes before local anesthetic injection, through the injection, and until completion of pulpotomy, assessed up to 35 minutes.
  Heart rate(beats per minute) was monitored using a pulse oximeter to evaluate the physiological stress response throughout treatment .Readings were recorded at predefined intervals. Increases in heart rate indicated heightened stress or discomfort during the procedure.
Oxygen saturation during dental procedures | From baseline measurement taken 5 minutes before local anesthetic injection, through the injection, and until completion of pulpotomy, assessed up to 35 minutes.
  Oxygen saturation (SpO₂, %) was monitored using a pulse oximeter to evaluate physiological stress response throughout treatment.Readings were recorded at predefined intervals. Decreases in SpO₂ indicated heightened stress or discomfort during the procedure.
Patient satisfaction with anesthesia technique | Immediately after the procedure
  Patient satisfaction was assessed using a structured questionnaire with two yes/no questions:
  1. Are you satisfied with the experience? (Yes/No)
  2. Would you like to have the same technique in future visits? (Yes/No) Responses were coded as binary outcomes (Yes = 1, No = 0). Higher total scores indicated greater patient satisfaction.
Parental satisfaction with anesthesia technique | Immediately after the procedure
  Parents rated their satisfaction using a Likert scale survey covering perceived child comfort and procedural experience. Scores ranged from 1 (very dissatisfied) to 5 (very satisfied). Higher scores reflected greater parental satisfaction with the anesthesia method used.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Wahab Nourallah, Prof, Principal Investigator — Faculty of Dentistry, Tishreen University; Sara Badr, PHD student, Principal Investigator — Faculty of Dentistry, Tishreen University
Locations (1):
- Faculty Of Dentistry ,Tishreen University, lattakia, Syria, Latakia, Syria

IPD SHARING:
Plan to Share IPD: No